CLINICAL TRIAL: NCT05638516
Title: Improving Mental Health in Youth and Lowering Risk for Obesity Through a Digital Preventative Product
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ksana Health (Industry)
Collaborators: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: OV-001
Record Dates: First submitted 2022-11-23; First posted 2022-12-06 (Actual); Last update posted 2023-05-18 (Actual); Status verified 2023-05

CONDITIONS: Mental Health Disorder; Obesity; Overweight
MeSH Terms: conditions — Mental Disorders; Obesity; Overweight

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vira Self-Care (Experimental): The Vira app is installed on the participant's phone. The app passively collects data from phone sensors (i.e., measures of physical activity, sleep patterns, mobility, and language patterns reflecting mood states and cognition) that are indicative of risk-relevant behavioral patterns and psychological states. It also so prompts users to answer a daily check in question. Mobile sensing data are processed to provide an automated assessment of the user's functioning. Users will be asked to use Vira for 12 weeks.
  The Vira app can be used as a standalone product. After an initial 10-day period, during which the app assesses the relationship between the user's patterns of behavior and their day-to-day variations in mental health and wellbeing using passive mobile sensing, the user is able to access a personalized behavior change goal that is support by in app information and functionality.
  Interventions: Behavioral: Vira mobile app intervention
- Vira + Coaching (Experimental): The Vira app can also be supported by a health coach. The health coach interacts with the user (via an instant messaging platform) and who also schedules just-in-time reminders (i.e., "nudges") to arrive in the user's phone at scheduled times to support their behavior change plan. The Vira Health Coach Platform therefore integrates mobile sensing, self-report assessment, and just-in-time nudges and notifications into the coach's workflow.
  Interventions: Behavioral: Vira mobile app intervention + coaching

INTERVENTIONS:
Behavioral: Vira mobile app intervention — The Vira app is installed on the participant's phone. The app passively collects data from phone sensors (i.e., measures of physical activity, sleep patterns, mobility, and language patterns reflecting mood states and cognition) that are indicative of risk-relevant behavioral patterns and psychological states. It also so prompts users to answer a daily check in question. Mobile sensing data are processed to provide an automated assessment of the user's functioning. Users will be asked to use Vira for 12 weeks.
  Arms: Vira Self-Care
Behavioral: Vira mobile app intervention + coaching — The Vira app can also be supported by a health coach. The health coach interacts with the user (via an instant messaging platform) and who also schedules just-in-time reminders (i.e., "nudges") to arrive in the user's phone at scheduled times to support their behavior change plan. The Vira Health Coach Platform therefore integrates mobile sensing, self-report assessment, and just-in-time nudges and notifications into the coach's workflow.
  Arms: Vira + Coaching

SUMMARY:
The goal of this study is to test the feasibility and utilization of a redesigned mobile app and health coaching platform (Vira) in youth (aged 18-25 years) with elevated depressive symptoms who are overweight/obese and/or self-report parental history of overweight/obesity.

Eligible participants will be randomly assigned to one of two groups: one group will use the Vira mobile app intervention with support from a health coach, and the other group will use the Vira mobile app intervention without coaching. Both groups will use the app for 12 weeks.

DETAILED DESCRIPTION:
The primary aim of this project is to examine the feasibility and utilization of a redesigned mobile app and health coaching platform (Vira) in a 2 x 2 (gender x condition) designed pilot study in a sample of 100 youth (18-25 years old) with (1) elevated depressive symptoms (PHQ-8 score ≥10) and (2) overweight/obesity (BMI ≥ 25 and/or reporting a parental history of overweight/obesity). The study will examine the feasibility and utilization of the mobile app intervention with coaching compared to that of the mobile app intervention without coaching.

This is an exploratory pilot study; therefore, no formal sample size calculation was conducted. It is anticipated that 1,000 individuals will be screened, of which 20% will be eligible, and that 50% of those eligible will agree to participate (final N = 100, 50 per arm).

ELIGIBILITY:
Inclusion Criteria:

* Age 18-25
* Live in the United States
* English fluency and literacy
* Have access to an Android or iOS device
* Elevated depressive symptoms (PHQ-8 score of 10 or above)
* Overweight (BMI of 25 or above) OR reporting a parental history of overweight or obesity

Exclusion Criteria:

* Previous participation in this study
* Major mental or physical illness that will interfere with completing intervention and/or assessment activities.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 73 (Actual)
Dates: Start 2022-11-07 (Actual); Primary Completion 2023-05-06 (Actual); Study Completion 2023-05-06 (Actual)

PRIMARY OUTCOMES:
Change in depressive symptoms | 12 weeks
  Pre- to post-intervention changes in depressive symptoms will be assessed by the Patient Health Questionnaire (PHQ-8) an 8-item participant-report measure for screening for depression and for establishing depression severity. The total score ranges from 0-24, with a higher score indicating greater depression symptom severity.
Number of active days in the Vira mobile app intervention and health coaching platform | 12 weeks
  To measure feasibility of implementation, the total number of active days using Vira during the study will be objectively collected via the Vira platform.
Number of features used | 12 weeks
  To measure feasibility of implementation, the total number of features used during the study will be objectively collected via the Vira platform.
Acceptability of the mobile app intervention | 12 weeks
  Acceptability of the mobile app intervention and health coaching platform will be assessed using 11 items adapted from the Technology Acceptance Model. Scores range from 11 to 77, with higher scores indicating greater acceptability.

CONTACTS AND LOCATIONS:
Overall Officials: Nick Allen, PhD, Principal Investigator — Ksana Health
Locations (1):
- Ksana Health, Eugene, Oregon, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Weiner LS, Crowley RN, Sheeber LB, Koegler FH, Davis JF, Wells M, Funkhouser CJ, Auerbach RP, Allen NB. Engagement, Acceptability, and Effectiveness of the Self-Care and Coach-Supported Versions of the Vira Digital Behavior Change Platform Among Young Adults at Risk for Depression and Obesity: Pilot Randomized Controlled Trial. JMIR Ment Health. 2024 Sep 19;11:e51366. doi: 10.2196/51366. PMID 39298763